CLINICAL TRIAL: NCT02084589
Title: A Comparison Study of Patient Controlled Epidural Analgesia (PCEA) With and Without Basal Infusion Using Ropivacaine 0,15% and Fentanyl μg/ml for Pain Relief in Labor, Assessment of Efficacy and Maternal Satisfaction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paraskevi Matsota (Other)
Responsible Party: Sponsor-Investigator, Paraskevi Matsota, MD, PhD, Attikon Hospital
Organization: Attikon Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101
Record Dates: First submitted 2014-03-05; First posted 2014-03-12 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Labor Pain
Keywords: PCEA, labor analgesia, background infusion, ropivacaine
MeSH Terms: conditions — Labor Pain | interventions — Fentanyl; Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- PCEA of continuous background infusion with demand dose (Active Comparator): PCEA with background infusion of 5 ml/h and demand dose of 5 ml with lockout 10 minutes, using ropivacaine 0,15% and fentanyl 2μg/ml.
  Interventions: Other: PCEA with basal infusion and demand dose using ropivacaine 0,15% and fentanyl 2μg/ml for pain relief in labor
- PCEA with demand dose only (Active Comparator): PCEA with demand dose of 5 ml with lockout 10 minutes, using ropivacaine 0,15% and fentanyl 2μg/ml.
  Interventions: Other: PCEA without basal infusion (demand only) using ropivacaine 0,15% and fentanyl 2μg/ml for pain relief in labor

INTERVENTIONS:
Other: PCEA with basal infusion and demand dose using ropivacaine 0,15% and fentanyl 2μg/ml for pain relief in labor
  Arms: PCEA of continuous background infusion with demand dose
Other: PCEA without basal infusion (demand only) using ropivacaine 0,15% and fentanyl 2μg/ml for pain relief in labor
  Arms: PCEA with demand dose only

SUMMARY:
This is a prospective, randomized, double blind study, in which a comparison of patient controlled epidural analgesia (PCEA) of continuous background infusion with demand dose and demand only, using ropivacaine 0,15% and fentanyl 2μg/ml for pain relief in labor, is being investigated. The purpose of the study is the assessment of the efficacy of labor analgesia and maternal satisfaction.

Written informed consent is obtained by all parturients. Non invasive monitor of blood pressure, heart rate, SpO2, ECG for the patient and a continuous monitoring of the fetal heart rate is being placed.

The participants are randomized in two groups, both receiving the same drug (ropivacaine 0,15% and fentanyl 2μg/ml). Group 0 receives demand dose of 5 ml with lockout of 10 minutes. Group 1 receives background infusion of 5 ml/h and demand dose of 5 ml with lockout 10 minutes.

All parturients have to be instructed to self administration of epidural bolus dose when they experience mild to moderate pain. Both parturient and anesthetist who conducts the study and treat breakthrough pain, are blind to group assignment.

After the last suture, total volume of epidural infusions of PCEA, total infused drug of PCEA pump, number of delivered PCEA boluses and manual rescue doses are being calculated. Time of delivery, mode of delivery, Apgar scores, and overall maternal satisfaction scores, neonate pH and Hct of the patient (ABGS), as well as possible need of newborn cardiopulmonary resuscitation are also recorded.

DETAILED DESCRIPTION:
This is a prospective, randomized, double blind study, in which a comparison of patient controlled epidural analgesia (PCEA) of continuous background infusion with demand dose and demand only, using ropivacaine 0,15% and fentanyl 2μg/ml for pain relief in labor, is being investigated. The purpose of the study is the assessment of the efficacy of labor analgesia and maternal satisfaction. Inclusion criteria include primigravidas or secundigravidas, 18 to 40 years old, ASA I or II, gestational age > 38 weeks, cervical dilatation ≥ 4 cm and request for epidural labor analgesia. Exclusion criteria are: patient's refusal to participate to the study, allergy to amino amide class of local anesthetics, contraindications to epidural analgesia, drug addiction or addiction to alcohol and administration of opioids in the last 3 hours before the initiation of labor epidural analgesia. Patients with history of clinical important cardiovascular, pulmonary, hepatic, neurological, psychiatric, metabolic or kidney disease are also excluded from the study.

After explaining the procedure to the parturient and the written consent is obtained, a preload of 500 ml of crystalloids is given intravenously. Non invasive monitor of blood pressure, heart rate, SpO2, ECG for the patient and a continuous monitoring of the fetal heart rate is being placed.

The insertion of the epidural catheter is performed at L2-L3, L3-L4 or L4-L5 interspace, in the sitting position, with 18G Touhy's needle using the loss of resistance to air technique to identify the epidural space. The catheter is inserted 4 cm into the epidural space and after aspiration for blood or cerebrospinal fluid is tested with 5 ml of drug containing ropivacaine 0,15% and fentanyl 2μg/ml. After 6 minutes and granted that verbal analogue score (VAS score) is ≥ 4, the PCEA pump is programmed.

The participants are randomized in two groups, both receiving the same drug (ropivacaine 0,15% and fentanyl 2μg/ml). Group 0 receives demand dose of 5 ml with lockout of 10 minutes. Group 1 receives background infusion of 5 ml/h and demand dose of 5 ml with lockout 10 minutes.

All parturients have to be instructed to self administration of epidural bolus dose when they experience mild to moderate pain (before the pain intensity becomes severe). Both parturient and anesthetist who conducts the study and treat breakthrough pain, are blind to group assignment. Breakthrough pain is defined as the manifestation of severe pain even with correct PCEA use, necessitating adjustment of analgesic regimen by the anesthesiologist during labor. In this case, the anesthetist controls the function of the epidural catheter and administrate a rescue dose of 5 ml of the drug and assess pain after 15 minutes. In case of VAS score more than 3 after 30 minutes and administration of two rescue doses, the parturient is withdrawn from the study and replaced by another parturient via randomization.

After the test dose and every 5 minutes for the first hour of labor the following parturients' parameters are collected; blood pressure, heart rate, SpO2, VAS score, level of sensory block and level of motor block (using the modified Bromage Scale), uterus contractions, oxytocin and possible side effects (nausea, vomiting, sedation, itch). Also, fetal heart rate is being recorded every five minutes. After the first hour and until the beginning of the second stage of labor the above parameters are monitored every 15 minutes, and from the second stage to the last suture every 5 minutes. Cervical dilatation is being recorded after every cervical examination performed by the obstetric team.

Maternal hypotension (defined as a systolic blood pressure (SPB) < 100 mmHg or a decrease of SBP of more than 20% from the baseline) is treated with left lateral position, administration of fluids and intravenous ephedrine (doses of 2,5 mg).

After the last suture, total volume of epidural infusions of PCEA, total infused drug of PCEA pump, number of delivered PCEA boluses and manual rescue doses are being calculated. Time of delivery, mode of delivery, Apgar scores, neonate pH and Hct of the patient (ABGS), as well as possible need of newborn cardiopulmonary resuscitation are also recorded. The epidural catheter is removed when the modified Bromage score is 6/6 and sensation is back to normal. At that point the overall maternal satisfaction is assessed.

The patient is under neurological exam for 24h (every 12 hours according to the protocol of our clinic).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 40 years,
2. ASA status I or II,
3. Primigravida or secundigravida
4. Gestational age > 38 weeks,
5. Cervical dilatation ≥ 4 cm,
6. Request for epidural labor analgesia

Exclusion Criteria:

1. Patients refusal to participate to the study
2. History of clinical important cardiovascular, pulmonary, hepatic, neurological, psychiatric, metabolic or kidney disease
3. Allergy to amino amide class of local anesthetics
4. Contraindications to epidural analgesia
5. Drug addiction or addiction to alcohol
6. Administration of opioids in the last 3 hours before the initiation of labor epidural analgesia
7. Use of chronic pain medications

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the total volume of epidural local anaesthetic (LA) administrated during labor. | Approximately 30 min (time of preloading) before the initiation of the epidural technique to 24 h after removal of the epidural catheter.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece